CLINICAL TRIAL: NCT06912737
Title: Development of a Group Emotion-Focused Behavioral Intervention for Diabetes Distress and Glycemic Management in Patients With T2D.
Brief Title: Group Emotion-Focused Behavioral Intervention for Diabetes Distress/A1c in T2D.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Emil Coccaro, George T. Harding Professor of Psychiatry & Behavioral Health, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024H0014; R01DK135948 (NIH)
Record Dates: First submitted 2024-12-27; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: T2DM (Type 2 Diabetes Mellitus)
Keywords: T2D; Diabetes Distress; HbA1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: Half of the study participants will be randomized to G-EFBI and half to G-WEHL.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Emotion Focused Behavioral Intervention (G-EFBI) (Experimental): Group EFBI (G-EFBI) is a 10-session, 75-minute, program aimed at assisting people with T2D to gain knowledge about emotions and improve their ability to regulate and manage their emotions. G-EFBI begins with discussions regarding the relationship between events, feelings, and behaviors/actions and how this relates to diabetes management. The intervention moves to teaching participants: (1) how to identify emotions and understand their purpose; (2) learn how identifying the physiological/behavioral pattern of their own emotions; (3) learn the importance of recognizing emotions in themselves and in others; (4) learn strategies aimed at helping them to better cope and manage their emotions; (5) learn to use specific emotional restructuring strategies (i.e., reframing, finding the evidence) to change their negative emotional responses to daily stressors and events as it relates to diabetes management.
  Interventions: Behavioral: Group Emotion Focused Behavioral Intervention (G-EFBI)
- G-WEHL (Active Comparator): To control for the effect of attention given to participants in G-EFBI that can result in psychosocial improvements, participants will be randomized to either G-EFBI or Group-With Every Heartbeat is Life (G-WEHL). G-WEHL is an educational intervention designed to increase awareness and prevention of cardiovascular disease. This intervention has ten 75-minute content sessions covering cardiovascular risk reduction in terms of diet, physical activity, and smoking cessation; the G-WEHL manual is provided in the Clinical Trials Section of this application; G-WEHL has no elements relevant to emotion regulation. The use of WEHL in this study is relevant because cardiovascular disease affects one-third of PWD, is a major cause of mortality (~ 50%), and impact (20-49%) on direct medical costs of T2D.
  Interventions: Behavioral: Group - With Every Heartbeat is Life (G-WEHL)

INTERVENTIONS:
Behavioral: Group Emotion Focused Behavioral Intervention (G-EFBI) — Group EFBI (G-EFBI) is aimed at assisting people with T2D to gain knowledge about emotions and improve their ability to regulate and manage their emotions.
  Arms: Group Emotion Focused Behavioral Intervention (G-EFBI)
Behavioral: Group - With Every Heartbeat is Life (G-WEHL) — G-WEHL is an educational intervention designed to increase awareness and prevention of cardiovascular disease.
  Arms: G-WEHL

SUMMARY:
T2D is a major public health problem and is currently the 7th leading cause of death in the US. Despite a range of efficacious treatments, less than 50% of patients achieve a glycemic target of A1c < 7.0%, suggesting that this is due to difficulty with following medical regimens to reduce A1C levels. While a range of factors have been identified in this regard, we posit that a barrier to treatment are broad difficulty with emotional regulation that are not diagnosis-specific but lead to Diabetes Distress (DD) and difficulty in coping with medical regimens, and other aspects of diabetes self-care, in the context of the psychosocial stressors associated with T2D. Extant data suggests that sub-optimal emotional regulation (experience of intense emotion and skill at regulating emotion) is related to elevated DD and A1c levels, and that an Emotion-Focused Behavioral Intervention (EFBI) can reduce both DD and A1c levels in PWD with T2D. In this project we seek to take our one-to-one intervention, now adapted to a group intervention (G-EFBI) and collect feasibility, acceptability, and preliminary efficacy data to determine if G-EFBI is a feasible, acceptable and, possibly, efficacious intervention compared to an "Attentional Control" intervention in PWD with T2D and elevated DD and A1c levels.

DETAILED DESCRIPTION:
This is an early-stage treatment development project proposing to conduct a modest randomized clinical trial of Group EFBI, vs. a Group Attentional Control Intervention, to collect feasibility, acceptability, and preliminary efficacy data in study participants with poorly controlled T2D (A1c > 7.5) and high Diabetes Distress Scale (DDS) scores (= or > 2 on any DDS subscale). This study will seek to study up to one hundred and twenty (120) study participants with T2D and elevated A1c and DDS scores will be recruited for about twelve (12) groups of seven to ten (7-10) to obtain feasibility, acceptability, and preliminary efficacy data. Participants will be randomized to ten 75-minute sessions of G-EFBI or of the Attentional Control Group Intervention, "With Every Heartbeat Is Life" (WEHL). WEHL is a psychoeducational intervention designed to increase awareness and prevention of cardiovascular disease and contains no ER related content. Study groups of patients with T2D will be recruited as above. This study will have 16 visits. Visit #1. Informed Consent and final assessment for study entry. Study participants must have a current A1c > 7.5%, a current DDS score > 2.0 on any DDS subscale, and be medically stable (e.g., without chronic renal failure). Assessments are listed below: 1. Glycemic Control. A1c using a DCA Vantage (Siemens) "point of contact" (POC) instrument. Blood (< 1 cc) is taken from a fingerstick. The total number of finger sticks in this study is four for a total blood collection volume of < 5 cc. 2. Diabetes Related Distress. Diabetes Distress Scale (DDS) 3. ER-Experience and ER-Skill. ER-Experience from the Affect Lability Scales (ALS); ER-Skill from the Trait-Meta-Mood (TMM) questionnaire. 4. Diabetes Self-Care and Engagement/Motivation. The Self-Care Inventory-Revised (SCI-R) and the Patient Activation Measure (PAM). 5. Depression, Anxiety, Stress, and Quality of Life (Q-LES-Q). State Depression/State Anxiety be assessed by PHQ-9 and GAD-7; Psychosocial stress assessed by the Perceived Stress Scale (PSS); Q-LES-Q will be assessed by Quality-of-Life Experience and Satisfaction. Visit #2: This is a 30-60 minute preparation session prior to the participant starting group intervention. Visit #3-7: Start G-EFBI or G-WEHL Sessions 1-5. Visit #8 (Mid-Point Assessment): A1c / DDS / AIM / ALS / TMM / SCI-R / PHQ-9 / GAD-7 / PSS / QOL. Visits 10-14: G-EFBI or G-WEHL Sessions 6-10. Visit #15 (End-Point Assessment): A1c / DDS / AIM / ALS / TMM / SCI-R / PHQ-9 / GAD-7 / PSS / Q-LES-Q. Visits #16 Post-Rx Assessment at Six Month F/U). Same as Visit #15.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults with documented diagnosis of T2D for at least one year.
2. Age > 18 years of age.
3. Diabetes Distress Scale score > 2.0 on any DDS subscale.
4. A1c > 7.5 (with hemoglobin in the normal range).
5. PHQ-9 Depression score < 15.
6. Stable medical co-morbid conditions.
7. Absence of a psychotic disorder or an intellectual disability.
8. Able to read English.
9. Able to give informed consent.

Exclusion Criteria:

1. Male and female adults with documented diagnosis of T2D for less than one year.
2. Age < 18 years of age.
3. Diabetes Distress Scale score < 2.0 on all DDS subscales.
4. A1c < 7.5 (with hemoglobin in the normal range).
5. PHQ-9 Depression score > 15.
6. Unstable medical co-morbid conditions (e.g., hospitalization in past three months).
7. Presence of a psychotic disorder or an intellectual disability.
8. Initiation of psychotherapy or pharmacotherapy for emotional issues within three months of study entry.
9. Unable to read English.
10. Unable to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Diabetes Distress Scale (DDS) | Week 0, Week 5, Week 10 and Month 6
  The Diabetes Distress Scale (DDS) will be used to assess psychological distress associated with the care and management of T2D; assessment of DD is critical for T2D intervention studies. The 17-item DDS has four subscales: regimen-related distress, emotional burden, physician distress, and interpersonal distress. Respondents have six options for each item ranging from "1" (not a problem) to "6" (a very serious problem). Mean Scores > 2.0 are at threshold for clinically meaningful DD.
HbA1c Level | Week 0, Week 5, Week 10 and Month 6
  A1c is measured at Visit #1 (Pre-Intervention) Visit #8 (Mid-Point), Visit #14 (After End of Intervention) and at Visit #15 (Six Month Follow-Up). A DCA Vantage (Siemens) "point of contact" (POC) instrument will be used for A1c levels. The research assistant will be trained in obtaining the fingerstick sample by the PI/Co-I (Drs. Coccaro and Joseph) and in how to operate the instrument. Our POC method displays a "unity" correlation with commercial assays (Roche Labs): r =.993 (p < .001) and bias of 0.03%.

SECONDARY OUTCOMES:
Emotion Regulation Skill (ER-Skill) | Week 0, Week 5, Week 10 and Month 6
  The "Clarity of Emotion" and "Repair of Emotion" scores from the Trait Meta-Mood (TMM) scale will constitute ER-Skill score.
Emotion Regulation Experience (ER-Exp) | Week 0, Week 5, Week 10 and Month 6
  The "Negative Emotional Intensity" score from the Affect Intensity Measure (AIM) and "Anxiety/Depression Lability" score from the Affect Lability Scales (ALS) will constitute the ER-Exp score.
Self-Care Inventory-Revised (SCI-R) | Week 0, Week 5, Week 10 and Month 6
  The Self-Care Inventory-Revised (SCI-R), included in our previous studies, will be used to assesses how well patients have followed self-care recommendations in the past month.
Patient Activation Measure (PAM) for Engagement/Motivation | Week 0, Week 5, Week 10 and Month 6
  The Patient Activation Measure (PAM), assessing skill/confidence for self-management will be used to assess engagement/motivation.
PHQ-9 for State Depression | Week 0, Week 5, Week 10 and Month 6
  State Depression will be assessed by commonly used PHQ-9 which is a nine-item screening assessment of current symptoms of depression.
GAD-7 for State Anxiety | Week 0, Week 5, Week 10 and Month 6
  State Anxiety will be assessed by GAD-7, a commonly used 7-item screening measure of state anxiety.
Perceived Stress Scale (PSS) for Perceived Psychosocial Stress | Week 0, Week 5, Week 10 and Month 6
  Perceived psychosocial stress will be assessed by the Perceived Stress Scale (Past Month). This is a ten item scale.
Quality of Life Experience and Satisfaction (Q-LES-Q) | Week 0, Week 5, Week 10 and Month 6
  Q=LES-Q is a 16-item QOL scale that assesses quality of life experience and satisfaction across several domains.
Assessment of Acceptance, Appropriateness, and Feasibility of Intervention. | Week 10 and Month 6
  Acceptability, Appropriateness, and Feasibility of Intervention (AAFI), as developed by Weiner et al. will be done at post-intervention (end of trial and six month follow-up). The AAFI comprises of three (3) four item Likert scale (1-5: strongly disagree to strongly agree) questionnaires with good internal (α's: 0.85 to 0.91) and test-retest (r=0.73 to 0.88), reliability known-groups validity, and sensitivity to change in both directions. These are Acceptability of Intervention Measure AIM), Intervention Appropriate Measure (IAM), and Feasibility of Intervention Measure (FIM).

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Demographic, clinical, and clinical trial data will be acquired from up to 120 individuals with Type 2 Diabetes. All data will be de-identified prior to receipt by the repository, but the information needed to generate a global unique identifier will be collected for each subject.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 1, 2030
Access Criteria: Any relevant health sciences investigator currently appointed at an academic institution.

DOCUMENTS (1):
  • Informed Consent Form (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT06912737/ICF_000.pdf